CLINICAL TRIAL: NCT00111683
Title: A Phase I/II Dose Escalation Study of MK0457 in Patients With Leukemia
Brief Title: MK0457 in Patients With Leukemia (0457-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-003; 2005_033
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Myelogenous Leukemia in Blast Crisis; Lymphocytic Leukemia, B Cell, Acute; Myelodysplastic Syndromes; Myelogenous Leukemia, Chronic
Keywords: Myelodysplastic Syndrome[Refractory Anemia with; Excess Blasts-1 or 2 (WHO Classification)]; Chronic Myelogenous Leukemia in blast crisis
MeSH Terms: conditions — Leukemia, Lymphoid; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — tozasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-0457 (Experimental): Participants receive MK-0457 as a continuous intravenous infusion (CIV) at assigned dose and duration
  Interventions: Drug: MK0457

INTERVENTIONS:
Drug: MK0457

SUMMARY:
In this study participants with relapsed/refractory leukemia will be given MK-0457 in sequential cohorts and with varying treatment duration to determine the maximum tolerated dose (MTD) for MK-0457.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Patients with relapsed/refractory acute myelogenous leukemia (AML), poor risk myelodysplastic syndrome (MDS), B-cell acute lymphocytic leukemia (ALL), myeloproliferative diseases, or chronic myelogenous leukemia (CML) in blast crisis

Part 2:

* Acute myelogenous leukemia (with FLT-3 mutation ), and myeloproliferative diseases only
* At least 2 weeks since the last cytotoxic therapy
* Acceptable renal and hepatic function
* Ambulatory, capable of all self-care, and out of bed for more than 50% of waking hours
* More than 2 months since autologous bone marrow or peripheral blood stem cell transplantation

Exclusion Criteria:

* Not fully recovered from previous anti-leukemia therapy
* Previous allogeneic bone marrow transplant
* Uncontrolled congestive heart failure
* Myocardial infarction within the last 3 months
* Active or uncontrolled infection
* Pregnancy or lactation
* Currently active second malignancy, other than non-melanoma skin cancer
* History of hepatitis B or C, known HIV positivity, or AIDS related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) | Part 1: up to 5 days, Part 2: up to 24 hours

SECONDARY OUTCOMES:
Hematological response rate to MK-0457 as a 5-day CIV infusion | At the end of each cycle (up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Giles FJ, Swords RT, Nagler A, Hochhaus A, Ottmann OG, Rizzieri DA, Talpaz M, Clark J, Watson P, Xiao A, Zhao B, Bergstrom D, Le Coutre PD, Freedman SJ, Cortes JE. MK-0457, an Aurora kinase and BCR-ABL inhibitor, is active in patients with BCR-ABL T315I leukemia. Leukemia. 2013 Jan;27(1):113-7. doi: 10.1038/leu.2012.186. Epub 2012 Jul 9. PMID 22772060